CLINICAL TRIAL: NCT05037695
Title: SGLT-2 Inhibitors in Prevention of Post-procedural Renal and Cardiovascular Complications aFter PCI Among Patients With Diabetes Mellitus and Coronary Artery Disease: a Prospective, Randomized, Pilot Study (SAFE-PCI)
Acronym: SAFE-PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Carlos Vicente Serrano Jr, MD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAFE-PCI
Record Dates: First submitted 2021-06-21; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease; Acute Kidney Injury
Keywords: PCI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Acute Kidney Injury | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, unblinded, randomized (1:1), single-center pilot study of 40 patients allocated to one of the treatment arms (OMT + empagliflozin or OMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- empagliflozin + OMT (Experimental): empagliflozin 25mg - Daily - at least 15 days before the PCI procedure OMT - Optimized Medical Therapy - conventional drug therapy with oral antidiabetics and/or insulin plus use of anti-platelet, anti-hypertensive and lipid-lowering agents necessary to obtain adequate values for pressure, lipid control and glycemia, in accordance with international guidelines and protocols. Strategies to reduce Contrast-induced acute kidney injury will be used in both study arms
  Interventions: Drug: empagliflozin 25 MG
- OMT (No Intervention): OMT - Optimized Medical Therapy - conventional drug therapy with oral antidiabetics and/or insulin plus use of anti-platelet, anti-hypertensive and lipid-lowering agents necessary to obtain adequate values for pressure, lipid control and glycemia, in accordance with international guidelines and protocols. Strategies to reduce Contrast-induced acute kidney injury will be used in both study arms

INTERVENTIONS:
Drug: empagliflozin 25 MG — empagliflozin 25mg - daily
  Arms: empagliflozin + OMT

SUMMARY:
Patients with type 2 diabetes mellitus (DM) have higher risk of major cardiovascular events (MACE) and renal disfunction. The Sodium-glucose cotransporter-2 inhibitors (iSGLT2) reduces hyperglycemia in patients with type 2 DM and have multiple metabolic effects, lowering primary composite cardiovascular outcomes and progression to renal failure. 25% of patients with Stable Ischemic Heart Disease (SIHD) undergoing PCI are diabetics being one of the most prevalent and important risk factors for the development of contrast induced nephropathy (CIN). The occurence of CIN is associated with higher rates of death, loss of renal function, necessity of dialysis and increase of health care costs. In this pilot study we sought to evaluate if the iSGLT2 would prevent periprocedural complications - such as periprocedural CIN and MI - in type 2 DM patients undergoing PCI through the assessment of renal and myocardial biomarkers

DETAILED DESCRIPTION:
* Prospective, unblinded, randomized (1:1), single-center pilot study of 40 patients allocated to one of the treatment arms (OMT + empaglifozin or OMT). Strategies to reduce Contrast-induced acute kidney injury will be used in both study arms
* The study population will be composed of patients with type II diabetes mellitus and coronary artery disease (CAD) suitable for PCI of one or more coronary vessels
* After discharge, all subjects will be clinically followed-up during hospitalization and for 30 days after PCI.
* Unless contra-indicated, all patients will receive intravenous hydration during 12 hours pre- and 12 hours post-PCI. Saline (NaCl 0.9%) infusion is recommended at a dose of 1 ml / kg body weight per hour and reduced to 0.5 ml/kg/h for those at high risk of volume overload (e.g. reduced left ventricular function or overt heart failure). All nephrotoxic drugs will be suspended at least 24 hours before the procedure.
* Operators will be strongly recommended to follow strict strategies to reduce the total volume of contrast for all patients
* All percutaneous procedures will be performed using non-ionic, low-osmolar or iso-osmolar, iodine-based contrast media
* The study groups will be compared according to the intention-to-treat principle. Categorical variables will be compared by Fisher's exact testing and continuous variables by Student's T testing. Time-dependent events will be estimated by the Kaplan-Meier method and compared by Hazards Cox modeling or log-rank test

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Type II Diabetes mellitus
* Finding of obstructive coronary artery disease (≥50% stenosis in major epicardial vessel) and clinical indication of percutaneous coronary intervention.(PCI)
* Participant is willing to comply with all aspects of the protocol, including adherence to the assigned strategy, medical therapy and follow-up visits
* Participant is willing to give written informed consent

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 30mL/min/1,73m2 or dialysis
* Inability to comply with the protocol
* Urgent need for PCI
* Acute coronary syndrome within the previous 30 days
* Use of iodinated contrast or other nephrotoxic agents < 7 days
* Angina after coronary bypass surgery
* Canadian Cardiovascular Society Class IV angina, including unprovoked rest angina
* Life expectancy less than the duration of the trial due to non-cardiovascular comorbidity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine values in pre-specified periods | Pre PCI
  Delta and area under curve
Serum creatinine values in pre-specified periods | Day 1
  Delta and area under curve
Serum creatinine values in pre-specified periods | Day 2
  Delta and area under curve
Serum creatinine values in pre-specified periods | Day 30
  Delta and area under curve
NGAL values in pre-specified periods | Pre PCI
  Delta and area under curve
NGAL values in pre-specified periods | Day 1
  Delta and area under curve
NGAL values in pre-specified periods | Day 2
  Delta and area under curve
NGAL values in pre-specified periods | Day 30
  Delta and area under curve

SECONDARY OUTCOMES:
Increase in serum creatinine ≥ 0.3 mg/dl or 50% from the baseline value, within 48 hours after the index procedure | 48 hours after PCI
  CI-AKI will be defined as an increase in serum creatinine ≥ 0.3 mg/dl or 50% from the baseline value, within 48 hours after the index procedure CI-AKI will be defined as an increase in serum creatinine ≥ 0.3 mg/dl or 50% from the baseline value, within 48 hours after the index procedure
Biomarkers elevation ≥10 upper reference limit (URL) for creatine kinase MB (CKMB) and/or ≥70 URL for troponin | 24 hours after PCI
  Periprocedural MI will be defined as biomarkers elevation ≥10 upper reference limit (URL) for creatine kinase MB (CKMB) and/or ≥70 URL for troponin
Occurrence of definite or probable stent thrombosis | Until 30 days
  Stent thrombosis will be defined as the occurrence of definite or probable stent thrombosis according to the Academic Research Consortium (ARC) criteria
Death From Cardiovascular Causes | Until 30 days
  Secondary Composite Outcome: Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, definite or probable stent thrombosis, stroke, bleeding (BARC 3-5) or death
Myocardial Infarction | Until 30 days
  Secondary Composite Outcome: Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, definite or probable stent thrombosis, stroke, bleeding (BARC 3-5) or death
Hospitalization for Unstable Angina | Until 30 days
  Secondary Composite Outcome: Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, definite or probable stent thrombosis, stroke, bleeding (BARC 3-5) or death
Stroke | Until 30 days
  Secondary Composite Outcome: Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, definite or probable stent thrombosis, stroke, bleeding (BARC 3-5) or death
Bleeding (BARC 3-5) | Until 30 days
  Secondary Composite Outcome: Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, definite or probable stent thrombosis, stroke, bleeding (BARC 3-5) or death
Death | Until 30 days
  Secondary Composite Outcome: Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, definite or probable stent thrombosis, stroke, bleeding (BARC 3-5) or death

CONTACTS AND LOCATIONS:
Overall Officials: Mateus P Feitosa, MD, Principal Investigator — Instituto do Coracao - HCFMUSP; Carlos V Serrano, MD, Study Director — Instituto do Coracao - HCFMUSP
Locations (1):
- Instituto do Coracao - HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehran R, Nikolsky E. Contrast-induced nephropathy: definition, epidemiology, and patients at risk. Kidney Int Suppl. 2006 Apr;(100):S11-5. doi: 10.1038/sj.ki.5000368. PMID 16612394
- [Background] Almendarez M, Gurm HS, Mariani J Jr, Montorfano M, Brilakis ES, Mehran R, Azzalini L. Procedural Strategies to Reduce the Incidence of Contrast-Induced Acute Kidney Injury During Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2019 Oct 14;12(19):1877-1888. doi: 10.1016/j.jcin.2019.04.055. Epub 2019 Sep 11. PMID 31521648
- [Background] Bahrainwala JZ, Leonberg-Yoo AK, Rudnick MR. Use of Radiocontrast Agents in CKD and ESRD. Semin Dial. 2017 Jul;30(4):290-304. doi: 10.1111/sdi.12593. Epub 2017 Apr 5. PMID 28382626
- [Background] Brenner BM, Cooper ME, de Zeeuw D, Keane WF, Mitch WE, Parving HH, Remuzzi G, Snapinn SM, Zhang Z, Shahinfar S; RENAAL Study Investigators. Effects of losartan on renal and cardiovascular outcomes in patients with type 2 diabetes and nephropathy. N Engl J Med. 2001 Sep 20;345(12):861-9. doi: 10.1056/NEJMoa011161. PMID 11565518
- [Background] Chang YK, Choi H, Jeong JY, Na KR, Lee KW, Lim BJ, Choi DE. Dapagliflozin, SGLT2 Inhibitor, Attenuates Renal Ischemia-Reperfusion Injury. PLoS One. 2016 Jul 8;11(7):e0158810. doi: 10.1371/journal.pone.0158810. eCollection 2016. PMID 27391020
- [Background] Das SR, Everett BM, Birtcher KK, Brown JM, Cefalu WT, Januzzi JL Jr, Kalyani RR, Kosiborod M, Magwire ML, Morris PB, Sperling LS. 2018 ACC Expert Consensus Decision Pathway on Novel Therapies for Cardiovascular Risk Reduction in Patients With Type 2 Diabetes and Atherosclerotic Cardiovascular Disease: A Report of the American College of Cardiology Task Force on Expert Consensus Decision Pathways. J Am Coll Cardiol. 2018 Dec 18;72(24):3200-3223. doi: 10.1016/j.jacc.2018.09.020. Epub 2018 Nov 26. No abstract available. PMID 30497881
- [Background] Donahoe SM, Stewart GC, McCabe CH, Mohanavelu S, Murphy SA, Cannon CP, Antman EM. Diabetes and mortality following acute coronary syndromes. JAMA. 2007 Aug 15;298(7):765-75. doi: 10.1001/jama.298.7.765. PMID 17699010
- [Background] Feres F, Costa RA, Siqueira D, Costa JR Jr, Chamie D, Staico R, Chaves AJ, Abizaid A, Marin-Neto JA, Rassi A Jr, Botelho R, Alves CMR, Saad JA, Mangione JA, Lemos PA, Quadros AS, Queiroga MAC, Cantarelli MJC, Figueira HR. DIRETRIZ DA SOCIEDADE BRASILEIRA DE CARDIOLOGIA E DA SOCIEDADE BRASILEIRA DE HEMODINAMICA E CARDIOLOGIA INTERVENCIONISTA SOBRE INTERVENCAO CORONARIA PERCUTANEA. Arq Bras Cardiol. 2017 Jun;109(1 Suppl 1):1-81. doi: 10.5935/abc.20170111. No abstract available. Portuguese. PMID 28792984
- [Background] Gilbert RE, Thorpe KE. Acute kidney injury with sodium-glucose co-transporter-2 inhibitors: A meta-analysis of cardiovascular outcome trials. Diabetes Obes Metab. 2019 Aug;21(8):1996-2000. doi: 10.1111/dom.13754. Epub 2019 May 24. PMID 31050116
- [Background] Haase M, Bellomo R, Devarajan P, Schlattmann P, Haase-Fielitz A; NGAL Meta-analysis Investigator Group. Accuracy of neutrophil gelatinase-associated lipocalin (NGAL) in diagnosis and prognosis in acute kidney injury: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Dec;54(6):1012-24. doi: 10.1053/j.ajkd.2009.07.020. Epub 2009 Oct 21. PMID 19850388
- [Background] Hueb W, Gersh BJ, Costa F, Lopes N, Soares PR, Dutra P, Jatene F, Pereira AC, Gois AF, Oliveira SA, Ramires JA. Impact of diabetes on five-year outcomes of patients with multivessel coronary artery disease. Ann Thorac Surg. 2007 Jan;83(1):93-9. doi: 10.1016/j.athoracsur.2006.08.050. PMID 17184637
- [Background] James MT, Ghali WA, Tonelli M, Faris P, Knudtson ML, Pannu N, Klarenbach SW, Manns BJ, Hemmelgarn BR. Acute kidney injury following coronary angiography is associated with a long-term decline in kidney function. Kidney Int. 2010 Oct;78(8):803-9. doi: 10.1038/ki.2010.258. Epub 2010 Aug 4. PMID 20686453
- [Background] Kidokoro K, Cherney DZI, Bozovic A, Nagasu H, Satoh M, Kanda E, Sasaki T, Kashihara N. Evaluation of Glomerular Hemodynamic Function by Empagliflozin in Diabetic Mice Using In Vivo Imaging. Circulation. 2019 Jul 23;140(4):303-315. doi: 10.1161/CIRCULATIONAHA.118.037418. Epub 2019 Feb 18. PMID 30773020
- [Background] Korner A, Eklof AC, Celsi G, Aperia A. Increased renal metabolism in diabetes. Mechanism and functional implications. Diabetes. 1994 May;43(5):629-33. doi: 10.2337/diab.43.5.629. PMID 8168637
- [Background] Lima EG, Hueb W, Garcia RM, Pereira AC, Soares PR, Favarato D, Garzillo CL, D'Oliveira Vieira R, Rezende PC, Takiuti M, Girardi P, Hueb AC, Ramires JA, Kalil Filho R. Impact of diabetes on 10-year outcomes of patients with multivessel coronary artery disease in the Medicine, Angioplasty, or Surgery Study II (MASS II) trial. Am Heart J. 2013 Aug;166(2):250-7. doi: 10.1016/j.ahj.2013.04.017. Epub 2013 Jun 15. PMID 23895807
- [Background] Ling W, Zhaohui N, Ben H, Leyi G, Jianping L, Huili D, Jiaqi Q. Urinary IL-18 and NGAL as early predictive biomarkers in contrast-induced nephropathy after coronary angiography. Nephron Clin Pract. 2008;108(3):c176-81. doi: 10.1159/000117814. Epub 2008 Feb 21. PMID 18287807
- [Background] Moussa ID, Klein LW, Shah B, Mehran R, Mack MJ, Brilakis ES, Reilly JP, Zoghbi G, Holper E, Stone GW. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Society for Cardiovascular Angiography and Interventions (SCAI). J Am Coll Cardiol. 2013 Oct 22;62(17):1563-70. doi: 10.1016/j.jacc.2013.08.720. PMID 24135581
- [Background] Ogurtsova K, da Rocha Fernandes JD, Huang Y, Linnenkamp U, Guariguata L, Cho NH, Cavan D, Shaw JE, Makaroff LE. IDF Diabetes Atlas: Global estimates for the prevalence of diabetes for 2015 and 2040. Diabetes Res Clin Pract. 2017 Jun;128:40-50. doi: 10.1016/j.diabres.2017.03.024. Epub 2017 Mar 31. PMID 28437734
- [Background] Ozkok S, Ozkok A. Contrast-induced acute kidney injury: A review of practical points. World J Nephrol. 2017 May 6;6(3):86-99. doi: 10.5527/wjn.v6.i3.86. PMID 28540198
- [Background] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Background] Ritz E, Orth SR. Nephropathy in patients with type 2 diabetes mellitus. N Engl J Med. 1999 Oct 7;341(15):1127-33. doi: 10.1056/NEJM199910073411506. No abstract available. PMID 10511612
- [Background] Solini A. Extra-glycaemic properties of empagliflozin. Diabetes Metab Res Rev. 2016 Mar;32(3):230-7. doi: 10.1002/dmrr.2666. Epub 2015 Jun 25. PMID 25994513
- [Background] Chu C, Lu YP, Yin L, Hocher B. The SGLT2 Inhibitor Empagliflozin Might Be a New Approach for the Prevention of Acute Kidney Injury. Kidney Blood Press Res. 2019;44(2):149-157. doi: 10.1159/000498963. Epub 2019 Apr 2. PMID 30939483
- [Background] Wanner C, Heerspink HJL, Zinman B, Inzucchi SE, Koitka-Weber A, Mattheus M, Hantel S, Woerle HJ, Broedl UC, von Eynatten M, Groop PH; EMPA-REG OUTCOME Investigators. Empagliflozin and Kidney Function Decline in Patients with Type 2 Diabetes: A Slope Analysis from the EMPA-REG OUTCOME Trial. J Am Soc Nephrol. 2018 Nov;29(11):2755-2769. doi: 10.1681/ASN.2018010103. Epub 2018 Oct 12. PMID 30314978
- [Background] Heyman SN, Khamaisi M, Rosen S, Rosenberger C, Abassi Z. Potential Hypoxic Renal Injury in Patients With Diabetes on SGLT2 Inhibitors: Caution Regarding Concomitant Use of NSAIDs and Iodinated Contrast Media. Diabetes Care. 2017 Apr;40(4):e40-e41. doi: 10.2337/dc16-2200. Epub 2017 Jan 27. No abstract available. PMID 28130255
- [Background] Tikkanen I, Narko K, Zeller C, Green A, Salsali A, Broedl UC, Woerle HJ; EMPA-REG BP Investigators. Empagliflozin reduces blood pressure in patients with type 2 diabetes and hypertension. Diabetes Care. 2015 Mar;38(3):420-8. doi: 10.2337/dc14-1096. Epub 2014 Sep 30. PMID 25271206
- [Background] Vallon V, Gerasimova M, Rose MA, Masuda T, Satriano J, Mayoux E, Koepsell H, Thomson SC, Rieg T. SGLT2 inhibitor empagliflozin reduces renal growth and albuminuria in proportion to hyperglycemia and prevents glomerular hyperfiltration in diabetic Akita mice. Am J Physiol Renal Physiol. 2014 Jan;306(2):F194-204. doi: 10.1152/ajprenal.00520.2013. Epub 2013 Nov 13. PMID 24226524
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Background] Weisbord SD, Gallagher M, Jneid H, Garcia S, Cass A, Thwin SS, Conner TA, Chertow GM, Bhatt DL, Shunk K, Parikh CR, McFalls EO, Brophy M, Ferguson R, Wu H, Androsenko M, Myles J, Kaufman J, Palevsky PM; PRESERVE Trial Group. Outcomes after Angiography with Sodium Bicarbonate and Acetylcysteine. N Engl J Med. 2018 Feb 15;378(7):603-614. doi: 10.1056/NEJMoa1710933. Epub 2017 Nov 12. PMID 29130810
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Derived] Feitosa MPM, Lima EG, Abizaid AAC, Mehran R, Lopes NHM, de Assis Fischer Ramos T, Hideo-Kajita A, Filho RK, Junior CVS. The safety of SGLT-2 inhibitors in diabetic patients submitted to elective percutaneous coronary intervention regarding kidney function: SAFE-PCI pilot study. Diabetol Metab Syndr. 2023 Jun 26;15(1):138. doi: 10.1186/s13098-023-01107-9. PMID 37365618